CLINICAL TRIAL: NCT03542006
Title: Brinzolamide for the Treatment of Chronic Central Serous Chorioretinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michaella Goldstein, Study Chair, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0647-17
Record Dates: First submitted 2017-10-28; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical brinzolamide (Experimental): Brinzolamide ophthalmic, given bd for 3 months
  Interventions: Drug: Brinzolamide Ophthalmic

INTERVENTIONS:
Drug: Brinzolamide Ophthalmic — Topical brinzolamide given bd for 3 months

SUMMARY:
Examine the efficacy of brinzolamide for the treatment of central serous chorioretinopathy

DETAILED DESCRIPTION:
Brinzolamide is a carbonic anhydrase inhibitor. Previously, carbonic anhydrase inhibitors have been shown to be effective for the treatment of macular edema when administered orally, also for central serous chorioretinopathy. However, this treatment carries the risk of severe side effects.

The goal of this study is to examine the efficacy of the topical form of treatment of carbonic anhydrase inhibitors in patients with chronic, non-resolving, central serous chorioretinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Central serous chorioretinopathy (CSC) affecting the fovea, non-resolving after 4 months of follow-up
* Optical coherence tomography (OCT) shows foveal subretinal fluid
* Fluorescein angiography and indocyanine green confirm the diagnosis

Exclusion Criteria:

* Any other ophthalmic condition that may lead to subretinal fluid
* Choroidal neovascularization
* Myopia > -6D
* Previous treatment for CSC in the past 6 months
* Known allergy to fluorescein or indocyanin green
* Known allergy for brinzolamide
* Pregnancy, breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in subretinal fluid (microns) | 6 months
  Change in subretinal fluid as measured by optical coherence tomography

SECONDARY OUTCOMES:
Change in ETDRS visual acuity (number of letters) | 6 months
  Change in visual acuity from baseline to last follow-up in ETDRS letters
Change in central macular thickness (microns) | 6 months
  Change in central macular thickness in microns from baseline to last follow-up
Change in choroidal thickness (microns) | 6 months
  Change in choroidal thickness in microns from baseline to last follow-up
Time for fluid resolution (days) | 6 months
  Time in days from baseline until fluid resolution, as measured on optical coherence tomography
Percentage of patients with fluid resolution | 6 months
  Percentage of patients with fluid resolution by last follow-up as seen on optical coherence tomography, out of all study participants
Quality of life assessment (using NEI-VFQ-25 questionnaires) | 6 months
  Quality of life score as assessed by standard questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Dinah Zur, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Iglicki Oftalmologia, Buenos Aires, Argentina
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No